CLINICAL TRIAL: NCT05970601
Title: Effects of Sodium Chloride or Its Substitute Salt Potassium Chloride on Vascular Function and Immune Response - a Randomized Controlled Trial
Brief Title: Effects of Sodium Chloride or Its Substitute Salt Potassium Chloride on Vascular Function
Acronym: ESCAPE-SALT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. med. Johannes Stegbauer (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Johannes Stegbauer, Assistant Professor, Heinrich-Heine University, Duesseldorf
Organization: Heinrich-Heine University, Duesseldorf (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2022-1844
Record Dates: First submitted 2023-07-08; First posted 2023-08-01 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Vascular Function; Healthy; Diabetes
Keywords: potassium chloride; sodium chloride; microcirculation
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- high salt group (Experimental): Intake of 9 g sodium chloride
  Interventions: Dietary Supplement: Soup
- low salt group (Active Comparator): Intake of 6 g sodium chloride
  Interventions: Dietary Supplement: Soup
- substitution group (Active Comparator): Intake of 6 g sodium chloride plus 3 g potassium chloride
  Interventions: Dietary Supplement: Soup

INTERVENTIONS:
Dietary Supplement: Soup — Intake of a single soup with different sodium chloride and potassium chloride content

SUMMARY:
This is a prospective, monocentric, randomized trial to investigate how sodium chloride or its substitute potassium chloride acutely affects vascular function by ingestion via a salted soup. Furthermore we want to get insights on the pathophysiology by analyzing metabolism and cell function in relation to vascular reaction.

DETAILED DESCRIPTION:
Some of the leading death causes in western countries are attributed to artheriosclerosis with its consequences especially cardiovascular events. Beside lifestyle risk factors such as physical inactivity, adipositas and stress, high dietary sodium intake is one of the easiest modifiable factors to reduce development and progession of artheriosclerosis. Unfortunately high sodium diet is one of the hallmarks of western diet. Epidemiologic and experimental data have provided compelling evidence that high salt and its induced elevation in bloodpressure is an important factor in the development and progression of cardiovascular disease, artheriosclerosis with its endorgan failure.

To analyze the reasons for the hazardous effects of high oral sodium chloride exposure on vascular damage and a possible protective mechanism by the salt substitute potassium chloride, we intend to conduct a single-center randomized trial (ESCAPE-SALT). We aim to measure vascular function by flow mediated dilation (FMD) and dynamic vessel analysis (DVA) of retinal mircocirculation. Participants will be divided into 3 groups. Each group will be served a soup with different salt content. The salt composition is as follows: soup A (9 g sodium chloride), soup B (6 g sodium chloride plus 3 g potassium chloride), and soup C (6 g sodium chloride). The effects on blood pressure, body composition markers, electrolytes, inflammatory and metabolic response, and vascular function are measured before, 4 and 24 h after ingestion of the soup. Furthermore we will investigate the underlying mechanism by performing metabolomic, transcriptomic and proteomic anyalysis.

ELIGIBILITY:
Inclusion Criteria:

* full-aged
* signed informed consent
* no dietary restrictions
* access to retina for microvascular measurement

Exclusion Criteria:

* age <18 y
* no retinal access for microvascular measurement
* known glaucoma
* antibiotic therapy within the last 4 weeks
* immunosuppressive Therapie within the last 4 weeks (e.g. glucocorticoids)
* s.p. malignancy
* unknown fever within the last 4 weeks
* salt wasting syndroms (e.g. renal tubular acidosis, Diabetes insipidus)
* chronic kidney disease stage 4-5
* known electrolyte disorder (e.g. hyperkalaemia, hypokalaemia, hypernatriaemia, hyponatriaema)
* no or rejected informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-08-09 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Effect of a single oral high-sodium chloride load or a partial substitution by potassium chloride on retinal vessel diameter and the flicker-light-induced retinal vessel dilatation. | Baseline, 4 hours, 24 hours
  Flicker-induced dilatation and diameter of fundus vessels will be measured via funduscopy in a static an dynamic analysis before, 4 hours and 24 hours after ingestion of a salty soup and the change between the timepoints will be analyzed. First the diameter of venoles and arterioles in µm and their ratio are measured in a standardized fundus picture. In a second step we will film the fundus during three flicker-light periods of 20 seconds and measure the dilatation in percent during the flicker period.
Effect of a single oral high-sodium chloride load or a partial substitution by potassium chloride on hypoxia-induced dilatation of brachial artery. | Baseline, 4 hours, 24 hours
  Flow mediated dilatation (FMD) as a marker for macrovascular function will be measured at baseline, 4 hours and 24 hours after ingestion of a salty soup. We will measure FMD by ultrasound based measurement of brachial artery diameter in mm before and after induced hypoxia for 5 minutes. The change of dilatation in percentage between the different timepoints will be analyzed.

SECONDARY OUTCOMES:
Effect of a single oral high-sodium chloride load or a partial substitution by potassium chloride on mitochondrial respiration capacity in PBMC. | Baseline, 4 hours, 24 hours
  Analysis of mitochondrial respiration capacity via seahorse technology in isolated PBMC from baseline, 4 and 24 hours after salt intake. The oxygen consumption rate (OCR) will be measured and the changes between the timepoints will be analyzed.
Effect of a single oral high-sodium chloride load or a partial substitution by potassium chloride on NO metabolism in serum and red blood cells. | Baseline, 4 hours, 24 hours
  We will measure the amount of nitrite and nitrate in red blood cells and serum by gas chemiluminescence at baseline, 4 and 24 hours after salt intake. The change between the three timepoints will be measured.
Effect of a single oral high-sodium chloride load or a partial substitution by potassium on metabolic profile in PBMC and plasma. | Baseline, 4 hours, 24 hours
  We will investigate the effect of a single oral high-sodium chloride load or a partial substitution by potassium on the metabolic profile in PBMCs and theplasma. The metabolites will be measured by liquid chromotagraphy and high resolution tandem mass spectrometry at baseline, 4 hours and 24 hours after salt intake. The difference between the timepoints will be analyzed.
Effect of a single oral high-sodium chloride load or a partial substitution by potassium on systemic inflammation markers. | Baseline, 4 hours, 24 hours
  Inflammatory markers such as cytokines will be meassured at baseline, 4 and 24 hours after salt intake by ELISA and OLINK. Changes of these markers between the three timepoints will be analyzed.

OTHER OUTCOMES:
Effect of a single oral high-sodium chloride load or a partial substitution by potassium chloride on fluid body composition. | Baseline, 4 hours, 24 hours
  Analysis of fluid body composition and intra- and extracellular water amount by bioimpendance monitoring at baseline, 4 and 24 hours after salt intake. The changes in body composition between the three timepoints will be measured.
Effect of a single oral high-sodium chloride load or a partial substitution by potassium chloride on blood pressure. | Baseline, 4 hours, 24 hours
  Analysis of blood pressure by automated office blood pressure device at baseline, 4 hours and 24 hours after salt intake. The changes in blood pressure between the three timepoints will be measured.
Effect of a single oral high-sodium chloride load or a partial substitution by potassium chloride on renin-angiotensine-aldosterone system. | Baseline, 4 hours, 24 hours
  Analysis of renin, angiotensine and aldosterone levels at baseline, 4 hours and 24 hours after salt intake, measurement will be done in the clinical routine laboratory and the difference between timepoints will be analyzed.
Effect of a single oral high-sodium chloride load or a partial substitution by potassium on fecal microbiome. | up to 48 hours before and after salt intake
  Analysis of the change of fecal microbiome composition in microbiology of probes before and after salt intake.
Effect of a single oral high-sodium chloride load or a partial substitution by potassium on metabolomics in stool. | up to 48 hours before and after salt intake
  Analysis of the change of metabolomics in stool and serum after salt intake using liquid chromotagraphy and high resolution tandem mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Stegbauer, MD, Principal Investigator — Heinrich-Heine University, Duesseldorf
Locations (1):
- University Hospital Düsseldorf, Heinrich Heine University, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No